CLINICAL TRIAL: NCT07403019
Title: A Prospective Cohort Study To Compare The Burden Of Medically Attended and Community RSV, hMPV, SARS-CoV-2 and Influenza LRTI In Infants And Children Under 5 Years Of Age and Adults (16-60 Years) In Rural India
Brief Title: Burden of Respiratory Viruses in India.
Status: Not yet recruiting | Type: Observational
Sponsor: MAHAN Trust (Other)
Responsible Party: Sponsor
Other Study IDs: MAHAN RSV 2025 1
Record Dates: First submitted 2026-02-04; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Pneumonia
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Biospecimen Retention: Samples With DNA — Nasopharyngeal swab collection
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort of 30 villages and 15 hospitals will be included.: We propose an active surveillance observational study in Melghat of a cohort of all newborns, infants and children under 5 years, and adults in age group of 16-60 years, for 36 months, of LRTI detected at home, primary health centers or hospitals in the catchment area of 30 villages under surveillance. The age range for the adult participants is 16-60 years.
  Interventions: Diagnostic Test: Nasopharyngeal swab for viral analysis

INTERVENTIONS:
Diagnostic Test: Nasopharyngeal swab for viral analysis — Active surveillance for LRTI cases in the community will be performed through weekly home visits by village health workers (VHWs) The VHWs are local women living in and accepted by the community. They have been trained using standard WHO materials, translated into Hindi. A nasopharyngeal swab will be obtained from children and adults (16-60 years) with non-severe, severe or very severe LRTI and those who die in 30 villages and 15 hospitals. A counselor is posted at every hospital and PHC who will capture every hospitalization of children under 5 and adults from the 30 villages, will identify any children from the 30 villages who visit the OPD with an LRTI and collect a swab from them. Children/adult with any lower respiratory illness will have a swab collected at admission and from any child/adult who dies. Samples (2000) will be tested for a panel of respiratory viruses first with a screening PCR(RSV, hMPV, SARS CoV 2 and Influenza) followed by subtyping when positive (RSV A

SUMMARY:
Trial Title: A Prospective Cohort Study To Compare The Burden Of Medically Attended and Community LRTI In Infants And Children Under 5 Years Of Age and adults (16-60 years) In India

Primary Objectives:

* To determine the population-based epidemiology, clinical features, and mortality of respiratory syncytial virus (RSV) lower respiratory tract illness (LRTI) in infants, children under 5, and adults (16-60 years) in rural India.
* To calculate the incidence of RSV LRTI classifications (non-severe, severe, very severe, hospitalization, and mortality) per 1,000 child/adult years of observation.

Secondary Objectives:

• To determine the population-based epidemiology of human metapneumovirus (hMPV), SARS-CoV-2, and influenza LRTI in the same cohort.

Study Design & Methodology:

* Type: Active surveillance, prospective longitudinal cohort study.
* Setting: 30 villages in the Melghat region of Maharashtra, India, characterized by high infant and adult mortality rates.
* Participants: All children under 5 years of age and adults aged 16-60 years residing in the study villages, including all newborns entering the cohort during the study period.
* Procedures: * Community Surveillance: Trained Village Health Workers (VHWs) will conduct weekly home visits to monitor respiratory health and identify potential LRTI cases.

  * Clinical Assessment: Supervisors will verify reported LRTI cases within 24 hours using standardized WHO classifications (non-severe, severe, and very severe pneumonia).
  * Medical Facility Monitoring: Hospital-based counselors will monitor all LRTI-related outpatient visits and hospitalizations from the study villages.
  * Sample Collection: Nasopharyngeal (NP) swabs will be collected from all identified LRTI cases (community and facility-based) and from any participant who dies within 15 days of an LRTI diagnosis.
  * Laboratory Testing: 2,000 samples will undergo real-time PCR screening and subtyping for RSV, hMPV, SARS-CoV-2, and influenza at the National Institute of Virology, Pune.
  * Mortality Investigation: For all participant deaths, a standardized verbal autopsy will be conducted to determine if LRTI was the cause of death.

Statistical Plan:

* Incidence rates and 95% confidence intervals will be calculated and severity category.
* Results will be stratified by age, sex, and socioeconomic status
* Multivariate analysis will be used Study Duration: 48 months total, including 36 months of active surveillance

DETAILED DESCRIPTION:
Study Title:

A Prospective Cohort Study To Compare The Burden Of Medically Attended and Community RSV, hMPV, SARS-CoV-2 and influenza LRTI In Infants And Children Under 5 Years Of Age and adults (16-60 years) In Rural India

Institution Name MAHAN Trust

Investigator Contact Information:

Dr. Ashish Satav Mahatma Gandhi Tribal Hospital, Karmgram, Utavali. Tahsil Dharni, District: Amaravati, Maharashtra. India pin: 444702 Phone : +919423118877 Email: drashish@mahantrust.org

Protocol ID MAHAN RSV 2025 1

Section #2- Core Protocol

2.1 Objectives & Hypotheses

2.1 Main objectives : Primary: To determine the population-based epidemiology of respiratory syncytial virus (RSV) lower respiratory tract illness (LRTI) in infants and children less than 5 years of age and adults, elderly people in rural India.

Secondary: To determine the population-based epidemiology of human metapneumovirus (hMPV), SARS-CoV-2 and influenza LRTI in infants and children less than 5 years of age and adults, elderly people in rural India, in relation to RSV.

2.1.1 Clinical hypotheses. This is primarily a descriptive observational study. However, we have proposed null hypotheses in the statistical methods, addressing each of the objectives and sub objectives

2.2 Background & Rationale, Significance of Selected Topic & Preliminary Data Respiratory syncytial virus (RSV) is the most common cause of infection of the upper and lower respiratory tract in infants and young children worldwide and is a major public health burden.1 2 It has been estimated that globally in 2019 there were 33.0 million episodes of RSV acute lower respiratory tract infections (LRTI) in children less than 5 years of age resulting in about 3.6 million hospitalizations, with 6.6 million episodes occurring in infants < 6 months of age and 1.4 million RSV associated ALRI hospitalizations 3. It was estimated that India bears a fifth of the global burden of illness (6.2 million episodes of RSV LRTI).3 Preliminary Data from our study the burden of RSV as a cause of mortality in rural infants and children under 2 years of age.

Results of Virology testing: In the 12 134 subjects, there were 5308 episodes of non-severe LRTI 2481 episodes of severe LRTIs and 1808 of very severe LRTIs. 4842 NP swabs were collected and tested by Real time RT-PCR for 16 respiratory viruses including RSV subtyping. During 2021 and 2022 additionally the samples were tested for SARS CoV 2. Out of 4842 almost 55% samples i.e., 2637 were positive for one or more respiratory viruses. RSV was detected in 740 cases (360 RSV A and 380 RSV B) followed by rhinovirus in 722 cases, PIV was detected in 345, Influenza 332, hMPV in 251, Adenovirus detected in 136. SARS CoV 2 was detected in 19 cases. RSV was detected in alternate year outbreaks with a dominance of RSV A or RSV B subtypes. In 2016 RSV A was predominantly in circulation where as in 2017 and 2018 RSV B was exclusively in circulation. In 2021 RSV A predominated. (Figure 1) RSV and hMPV alternate and Influenza occurs annually.

RSV Mortality: Fifteen of 16(94%) children with RSV died of LRTI, 14 in the community and 1 in the hospital. The case fatality ratios for severe RSV LRI in the first 6 months of life were 3/52(7.1%) and 1/36(2.8%) in the community and hospital respectively. Of those with very severe LRTI in the community, 17.6% died. There were no very severe RSV LRTI hospital deaths. The adjusted RSV LRTI mortality rates ranged from 1.0 - 3.0/1000 child years (CY) overall, and 2.0 - 6.1/1000 CY, accounting for 20% of the LRTI deaths and 10% of the post neonatal infant mortality.4

2.3 Study Design Melghat is a hilly, forested area spread over >4000 km2 in Maharashtra state, Central India, with population of 2,80,000 scattered over 320 villages, distributed in 2 blocks. The government primary health care delivery is through sub-center with paramedical workers for 2-5 villages, a Primary Health Center (PHC) with a doctor and nurses for every 30 villages, a rural sub-district hospital (RH) and 2 district hospitals 1 for mother and children and the other for adults. MAHAN hospital, where the study is based is a charitable trust hospital that provides free or low-cost care to the community.

We propose an active surveillance observational study in Melghat of a cohort of all newborns, infants and children under 5 years, and adults in age group of 16-60 years, for 36 months, of LRTI detected at home, primary health centers or hospitals in the catchment area of 30 villages under surveillance. Active surveillance for LRTI cases in the community will be performed through weekly home visits by village health workers (VHWs) The VHWs are local women living in and accepted by the community. They have been trained using standard WHO materials, translated into Hindi with a refresher course every 6 months. A nasopharyngeal swab will be obtained from children and adults (16-60 years) with non-severe, severe or very severe LRTI and those who die. A counselor is posted at every hospital and PHC who will capture every hospitalization of children under 5 and adults from the 30 villages, will identify any children from the 30 villages who visit the OPD with an LRTI and collect a swab from them. Children/adult with any lower respiratory illness will have a swab collected at admission and from any child/adult who dies. Samples (2000) will be tested for a panel of respiratory viruses first with a screening PCR(RSV, hMPV, SARS CoV 2 and Influenza) followed by subtyping when positive (RSV A and RSV B; hMPV A and hMPV B; Influenza A H1N1 pdm2009, H3N2 and Influenza B and SARS CoV 2 ) at the National Institute of Virology, Pune.

2.7 Study Procedures Study Population: At the start of the study All children under the age of five years and adults (16-60 years) will be recruited for prospective observation for LRTI, after obtaining informed consent from the parent/caretaker. Subsequently using pregnancy monitoring, all parents of live-born neonates will be approached for consent to follow-up their children for the next 3 years. Subjects will be followed until they reach the age of 5 years or 60 years, migrate permanently out of the 30 villages, withdrew consent, or expire.

Health worker training:

All VHWs, and their supervisors and health center/hospital based counselors will be re-trained using a modified World Health Organization (WHO) methodology, in the recognition of WHO defined Pneumonia5, and its recording on paper case report forms as well as how to collect nasopharyngeal (NP) swabs in infants and children, and adults (16-60 years).

Subject monitoring in the community:

Our experience is that VHWs develop a keen rapport with the families who they follow with weekly home visits, specifically following the respiratory health of the subjects. Any child or adult with an LRTI, will have a NP swab collected for pathogen detection. Treatment will follow Govt. of Maharashtra guidelines that permits VHW's to prescribe amoxicillin for pneumonia/ within 24 hours of the assessment, supervisors will visit the subject and conduct a respiratory assessment as well. All subjects with LRTI who are hospitalized, will be followed up at home one and two weeks later. (Follow up form) VHWs are also informed of community deaths and, after grief counseling is offered to the family, either by a supervisor or local trained traditional healers or nurses, with informed consent, NP swabs will be obtained from the deceased child whenever feasible. (the community is used to this)

Subject monitoring in the health centers and hospitals:

Counselors working in the 14 government facilities will monitor the outpatient and conduct a daily census of all new admissions, and after obtaining informed consent, (from children and adults from the 30 villages) will administer a short questionnaire and collect a NP sample from children (0-5 years) and adults (16-60 years) with LRTI or sepsis, as well as all who die. (if they have not been already collected by the VHW in the village) for an acute illness visit . Total samples to be collected 2000.

Nasopharyngeal swab collection and sample processing:

NP swabs will be collected using flocked swabs and transported in viral transport medium to MAHAN hospital where they will be stored at 4-80C. Batches are transported to the ICMR -National Institute of Virology Pune for pathogen testing. The samples will be tested in a 2-step manner (screening and subtyping) as outlined previously by real time PCR using standardized protocols6,7.

Verbal Autopsy:

A supervisor and a VHW from the community will conduct a verbal autopsy (VA) within 2 weeks of the death. The VA uses standardized Indian government protocols modified for use in Maharashtra incorporating local terminology8,9. The narratives are read by two independent trained physicians, and where there is discordance, a third Senior pediatrician adjudicates the difference.

All pathogen testing is done at India's premier virology Institute, National Institute of Virology, Pune.

2.8 Study duration and study timelines

The study will proceed in four major phases over a 4-year implementation period:

2.10Statistical Analysis and Sample Size Justification Statistical Analysis Plan All data will be entered into a RedCap database and exported for analysis. All statistical analyses will be done by the Biostatistician Dr Raje, who is part of the study team,

Statistical methods The demographic and socio-economic status of each subject included in the cohort will be summarized according to scale of measurement. Continuous variables with be expressed in terms of mean and standard deviation, while categorical variables will be summarized in terms of frequencies and percentages.

Primary objective

1. To prospectively determine the burden (clinical features and mortality) of RSV LRTI in a cohort of infants and children under 5 and adults (16-60 years) in 30 villages, over 3 years, and all newborns entering the cohort during the 3 years of the study.
2. To determine the incidence (per 1000 child years/adult years of observation) of the following classifications of RSV LRTI, using the WHO classification of disease: non-severe pneumonia, severe pneumonia, very severe pneumonia, RSV hospitalization, RSV mortality.
3. To evaluate the RSV subgroup specific (RSV A and RSV B) burden of illness and to compare severity based on subgroups.

Power/Sample Size:

We plan to recruit a cohort of 22,121 individuals, comprising:

* 2,726 children aged 0-5 years (U5C)
* 19,395 adults aged 16-60 years, These sample sizes are powered to detect statistically significant differences (α = 0.05, power = 80%) in virus-specific respiratory disease incidence between subgroups (e.g., age, nutrition status, tribal subpopulation) and to analyse long-term sequelae patterns in RSV-positive vs. RSV-negative individuals using lung function tests.

2.16 Plan for Policy Translation Proactive dissemination and policy translation plan will be implemented.

* Continuous Stakeholder Engagement:
* Evidence-Based Advocacy:
* Targeted Dissemination of Findings:

  * Policy Briefs:
  * Academic Publications:
  * Conferences and Meetings:
  * Public interest litigation to courts.
* Public and Community-Level Communication:

2.17 Local Stakeholder Engagement Strategy for Engaging Local Stakeholders To maximize the study's relevance, impact, and long-term sustainability, this plan outlines a dedicated strategy for the early and continuous engagement of local health authorities and policymakers.

1. Initial Partnership Building and Alignment
2. Formation of a Stakeholder Advisory Group
3. Regular and Transparent Communication
4. Integration with Existing Health Systems o

ELIGIBILITY:
Inclusion Criteria:

* All children (0-5 years) and adults (16-60 years) from 30 villlages and 15 hospitals will be included in the study who are sufffering from pneumonia or who died. Informed written consent from parents, patients and spouse or children in necessary

Exclusion Criteria:

* All other healthy people from the study area will be excluded or who donot give informed written consent will be excluded.

Ages: 1 Minute to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study is based on a poor rural population of Melghat, Amaravati district of Maharashtra in India, where all of the participants are of Indian origin/descent. Since India is the single most important country contributing to the burden of morbidity and mortality of respiratory illness globally, and most of this occurs in parts of rural India where infant mortality and adult mortality still remains high, this population is the exact population where studies on the viral epidemiology and burden need to be conducted. Hence this population though not diverse, is a highly relevant population whether burden of disease occurs, but is really unstudied till our preceding study referenced in the text.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2030-03-31 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
To determine the population-based epidemiology of respiratory syncytial virus (RSV) lower respiratory tract illness (LRTI) in infants and children less than 5 years of age and adults, elderly people in rural India. | 48 months
  1. To prospectively determine the clinical features and mortality from RSV lower respiratory tract illness in a cohort of infants and children under 5 years and adults, elderly people in 30 villages, over 3 years, and all newborns entering the cohort during the 3 years of the study.
  2. To determine the incidence (per 1000 child years and adults, elderly people of observation) of the following classifications of RSV LRTI, using the WHO classification of disease: non-severe pneumonia, severe pneumonia, very severe pneumonia, RSV hospitalization, RSV mortality.
  3. To evaluate the RSV subgroup specific (RSV A and RSV B) burden of illness and to compare severity and incidence based on subgrouping.

CONTACTS AND LOCATIONS:
Overall Officials: Ashish R Satav, MBBS. MD, Principal Investigator — MAHAN Trust
Locations (1):
- Mahatma Gandhi Tribal Hospital Karmgram Utavali Dharni Amaravati, Amravati, Maharashtra, India

IPD SHARING:
Plan to Share IPD: No
Indian government donot permit to share the individual participant data.

REFERENCES:
- [Background] Collier F, Choain MC, Letombe B, Pagniez I, Gauthier A. [FSH in ovulation induction from theory to practice]. Contracept Fertil Sex. 1995 May;23(5):291-301. No abstract available. French. PMID 7613574
- [Background] Li Y, Wang X, Blau DM, Caballero MT, Feikin DR, Gill CJ, Madhi SA, Omer SB, Simoes EAF, Campbell H, Pariente AB, Bardach D, Bassat Q, Casalegno JS, Chakhunashvili G, Crawford N, Danilenko D, Do LAH, Echavarria M, Gentile A, Gordon A, Heikkinen T, Huang QS, Jullien S, Krishnan A, Lopez EL, Markic J, Mira-Iglesias A, Moore HC, Moyes J, Mwananyanda L, Nokes DJ, Noordeen F, Obodai E, Palani N, Romero C, Salimi V, Satav A, Seo E, Shchomak Z, Singleton R, Stolyarov K, Stoszek SK, von Gottberg A, Wurzel D, Yoshida LM, Yung CF, Zar HJ; Respiratory Virus Global Epidemiology Network; Nair H; RESCEU investigators. Global, regional, and national disease burden estimates of acute lower respiratory infections due to respiratory syncytial virus in children younger than 5 years in 2019: a systematic analysis. Lancet. 2022 May 28;399(10340):2047-2064. doi: 10.1016/S0140-6736(22)00478-0. Epub 2022 May 19. PMID 35598608
- [Background] Simoes EAF, Dani V, Potdar V, Crow R, Satav S, Chadha MS, Hessong D, Carosone-Link P, Palaskar S, Satav A. Mortality From Respiratory Syncytial Virus in Children Under 2 Years of Age: A Prospective Community Cohort Study in Rural Maharashtra, India. Clin Infect Dis. 2021 Sep 2;73(Suppl_3):S193-S202. doi: 10.1093/cid/ciab481. PMID 34472578
- [Background] Madhi SA, Polack FP, Piedra PA, Munoz FM, Trenholme AA, Simoes EAF, Swamy GK, Agrawal S, Ahmed K, August A, Baqui AH, Calvert A, Chen J, Cho I, Cotton MF, Cutland CL, Englund JA, Fix A, Gonik B, Hammitt L, Heath PT, de Jesus JN, Jones CE, Khalil A, Kimberlin DW, Libster R, Llapur CJ, Lucero M, Perez Marc G, Marshall HS, Masenya MS, Martinon-Torres F, Meece JK, Nolan TM, Osman A, Perrett KP, Plested JS, Richmond PC, Snape MD, Shakib JH, Shinde V, Stoney T, Thomas DN, Tita AT, Varner MW, Vatish M, Vrbicky K, Wen J, Zaman K, Zar HJ, Glenn GM, Fries LF; Prepare Study Group. Respiratory Syncytial Virus Vaccination during Pregnancy and Effects in Infants. N Engl J Med. 2020 Jul 30;383(5):426-439. doi: 10.1056/NEJMoa1908380. PMID 32726529
- [Background] Simoes EA, Mutyara K, Soh S, Agustian D, Hibberd ML, Kartasasmita CB. The epidemiology of respiratory syncytial virus lower respiratory tract infections in children less than 5 years of age in Indonesia. Pediatr Infect Dis J. 2011 Sep;30(9):778-84. doi: 10.1097/INF.0b013e318218ab9e. PMID 21487330
- [Background] Satav A, Crow R, Potdar V, Dani V, Satav S, Chadha M, Hessong D, Carosone-Link P, Palaskar S, Simoes EAF. The Burden of Respiratory Syncytial Virus in Children Under 2 Years of Age in a Rural Community in Maharashtra, India. Clin Infect Dis. 2021 Sep 2;73(Suppl_3):S238-S247. doi: 10.1093/cid/ciab508. PMID 34472575
- See also: A Prospective Cohort Study To Compare The Burden Of Medically Attended and Community RSV, hMPV, SARS-CoV-2 and influenza LRTI In Infants And Children Under 5 Years Of Age and adults (16-60 years) In Rural India — https://www.mahantrust.org/
- Available data/document: Study Protocol — https://www.mahantrust.org/copy-of-research-papers